CLINICAL TRIAL: NCT06677957
Title: A Phase I, Open-Label, Two-Period, One-Sequence, Crossover Study in Healthy Subjects to Evaluate the Clinical Drug-Drug Interaction of Divarasib With Probe Substrates of P-Glycoprotein (Digoxin) and Breast Cancer Resistance Protein (Rosuvastatin)
Brief Title: A Clinical Trial to Investigate the Clinical Drug-Drug Interaction of Divarasib With Probe Substrates of P-Glycoprotein and Breast Cancer Resistance Protein in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GP45712
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Digoxin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Participants will receive a single oral dose of Digoxin and Rosuvastatin drug cocktail.
  Interventions: Drug: Digoxin; Drug: Rosuvastatin
- Treatment B (Experimental): Participants will receive a single dose of Digoxin and Rosuvastatin drug cocktail administered 2 hours after the Divarasib dose on Day 5.
  Interventions: Drug: Digoxin; Drug: Divarasib; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Digoxin — Digoxin will be administered together with Rosuvastatin as a drug cocktail as specified for the respective period
Drug: Divarasib — Divarasib will be administered in combination with Digoxin and Rosuvastatin as specified for the respective period
  Arms: Treatment B
Drug: Rosuvastatin — Rosuvastatin will be administered together with Digoxin as a drug cocktail as specified for the respective period

SUMMARY:
This is a Phase 1, open-label, two-period, one-sequence, crossover drug-drug interaction study to assess the P-gp and BCRP inhibition potential of divarasib using digoxin and rosuvastatin as probe substrates, respectively, in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-childbearing potential
* Within body mass index (BMI) range of 18.0 to 32.0 kg/m2, inclusive

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal (GI), neurological, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator
* Poor peripheral venous access

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Digoxin and Rosuvastatin | Day 1 of Period 1 and Day 5 of Period 2
Area Under the Plasma Concentration-Time Curve from Hour 0 to the Last Measurable Concentration (AUC0-t) of Digoxin and Rosuvastatin | Day 1 of Period 1 and Day 5 of Period 2
Area Under the Plasma Concentration-Time Curve (AUC0-inf) of Digoxin and Rosuvastatin | Day 1 of Period 1 and Day 5 of Period 2
Time to Cmax (Tmax) of Digoxin and Rosuvastatin | Day 1 of Period 1 and Day 5 of Period 2

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | From Day 1 until end of study participation (approximately 2 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Daytona Beach Clinical Rsch Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No